CLINICAL TRIAL: NCT00838110
Title: A Phase 3, Multi-Center, Randomized, Double-Blind Placebo-Controlled Study To Evaluate The Safety And Tolerability Of Dimebon (PF-01913539) For Up To 26-Weeks In Patients With Mild To Moderate Alzheimer's Disease
Brief Title: A Phase 3 Study To Evaluate The Safety And Tolerability Of Dimebon Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1451027
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Dimebon; Safety; Tolerability
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dimebon 20 mg TID (Cohort 1) (Experimental)
  Interventions: Drug: Dimebon
- Placebo TID (Cohort 1) (Placebo Comparator)
  Interventions: Drug: Placebo
- Dimebon 20 mg TID (Cohort 2) (Experimental)
  Interventions: Drug: Dimebon
- Placebo TID (Cohort 2) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimebon — 10 mg TID for week 1 followed by 20 mg TID through Week 26
  Arms: Dimebon 20 mg TID (Cohort 1)
Drug: Placebo — 10 mg TID for week 1 followed by 20 mg TID through Week 26
  Arms: Placebo TID (Cohort 1)
Drug: Dimebon — 10 mg TID for week 1 followed by 20 mg TID through Week 12
  Arms: Dimebon 20 mg TID (Cohort 2)
Drug: Placebo — 20 mg matched Placebo (Cohort 2) 10 mg TID for week 1 followed by 20 mg TID through Week 12
  Arms: Placebo TID (Cohort 2)

SUMMARY:
This is a multi-center, randomized, double-blind placebo-controlled safety study conducted in 2 study cohorts. In Cohort 1, subjects with Alzheimer's disease (n=250) will receive Dimebon 20 mg or placebo TID for 26 weeks. In Cohort 2 AD subjects (n=500) will be treated with Dimebon 20 mg or placebo TID for 12 weeks After completion of the randomized portion of the study, subjects in both Cohorts will have the opportunity to enroll in a Dimebon open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease.
* MMSE 12-26 inclusive.
* If on existing anti-dementia therapy, have been on a stable dose of anti-dementia therapy (cholinesterase inhibitors and/or memantine) for at least 60 days prior to dosing in study.
* If not taking existing anti-dementia therapy, have not received therapy with cholinesterase inhibitors and/or memantine within 60 days prior to dosing in this study.

Exclusion Criteria:

* Have major structural brain disease (e.g., ischemic infarcts, subdural hematoma, hemorrhage, hydrocephalus, brain tumors, multiple subcortical ischemic lesions, or a single lesion in a critical region [e.g., thalamus, hippocampus]).
* Have any major medical illness or unstable medical condition within six months of screening that may interfere with the patient's ability to comply with study procedures and abide by study restrictions.
* Have not been on a stable dose of anti-dementia therapy for at least 60 days prior to dosing or intend to start anti-dementia therapy during the double blind portion of the study.
* Reside in a nursing home or assisted care facility with need for 24-hour care and supervision.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (108):
- United States (85):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Northport, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Pueblo, Colorado
  - Pfizer Investigational Site, Hockessin, Delaware
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Fort Walton Beach, Florida
  - Pfizer Investigational Site, Fruitland Park, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Plant City, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Burr Ridge, Illinois
  - Pfizer Investigational Site, Elk Grove Village, Illinois
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Greenfield, Indiana
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, West Yarmouth, Massachusetts
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Great Falls, Montana
  - Pfizer Investigational Site, Eatontown, New Jersey
  - Pfizer Investigational Site, Oakhurst, New Jersey
  - Pfizer Investigational Site, Toms River, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Grove City, Pennsylvania
  - Pfizer Investigational Site, Indiana, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Scotland, Pennsylvania
  - Pfizer Investigational Site, Upper Saint Clair, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Murrells Inlet, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Carrollton, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Grand Prairie, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Williamsburg, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Charleston, West Virginia
  - Pfizer Investigational Site, La Crosse, Wisconsin
- Canada (19):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Medicine Hat, Alberta
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Pfizer Investigational Site, Kentville, Nova Scotia
  - Pfizer Investigational Site, Pictou, Nova Scotia
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint-Jean-sur-Richelieu, Quebec
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Puerto Rico (4):
  - Pfizer Investigational Site, Cayey, PR
  - Pfizer Investigational Site, Rio Piedras, PR
  - Pfizer Investigational Site, San Juan, PR
  - Pfizer Investigational Site, Cidra

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451027

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimebon (Cohort 1): Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day up to Week 26.
- Placebo (Cohort 1): Placebo tablet matched to 10 mg of dimebon (latrepirdine) tablet orally three times a day for 1 week (titration period), followed by placebo tablet matched to 20 mg dimebon (latrepirdine) tablet orally three times a day up to Week 26.
- Dimebon (Cohort 2): Dimebon (latrepirdine) 10 mg tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day up to Week 12.
- Placebo (Cohort 2): Placebo tablet matched to 10 mg of dimebon (latrepirdine) tablet orally three times a day for 1 week (titration period), followed by placebo tablet matched to 20 mg dimebon (latrepirdine) tablet orally three times a day up to Week 12.
Period: Overall Study
Arm/Group | Dimebon (Cohort 1) | Placebo (Cohort 1) | Dimebon (Cohort 2) | Placebo (Cohort 2)
Started | 127 | 128 | 243 | 244
Treated | 127 | 127 | 243 | 244
Completed | 105 | 106 | 226 | 226
Not Completed | 22 | 22 | 17 | 18
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Adverse Event | 11 | 10 | 8 | 7
Not completed — Withdrawal by Subject | 5 | 6 | 3 | 4
Not completed — Other | 3 | 3 | 3 | 2
Not completed — Protocol Violation | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Did not meet eligibility criteria | 0 | 0 | 1 | 2
Not completed — Randomized but not treated | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dimebon: Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day up to Week 26 for cohort 1 and up to Week 12 for cohort 2.
- Placebo: Placebo tablet matched to 10 mg of dimebon (latrepirdine) tablet orally three times a day for 1 week (titration period), followed by placebo tablet matched to 20 mg dimebon (latrepirdine) tablet orally three times a day up to Week 26 for cohort 1 and up to Week 12 for cohort 2.
- Total: Total of all reporting groups
Arm/Group | Dimebon | Placebo | Total
Number analyzed (Participants) | 370 | 371 | 741
Age, Customized [Number; unit: Participants]
  50 to 59 years | 24 | 13 | 37
  60 to 69 years | 50 | 63 | 113
  70 to 79 years | 155 | 154 | 309
  80 to 85 years | 109 | 103 | 212
  Greater than 85 years | 32 | 38 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 198 | 390
  Male | 178 | 173 | 351

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Vital Signs in Cohort 1
Description: Abnormal clinically significant vital signs included absolute systolic blood pressure (BP) values: less than (<) 90 millimeter of mercury (mmHg), maximum increase or decrease of greater than or equal to (>=) 30 mmHg from baseline; absolute diastolic BP value: <50 mmHg, maximum increase or decrease of >=20 mmHg from baseline; absolute heart rate values: >120 beats per minute (bpm).
Time Frame: Baseline up to Week 30 (follow-up)
Population: Cohort 1 analysis set included all those participants in the safety analysis set (SAS) (all participants who receive at least one dose of study medication, including partial doses) who were randomized into cohort 1 of the study. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 1) | Placebo (Cohort 1)
Number analyzed (Participants) | 127 | 127
percentage of participants
  Systolic BP (<90 mmHg) (n=127,127) | 0.8 | 1.6
  Increase in systolic BP (>=30 mmHg) (n=126,124) | 9.5 | 10.5
  Decrease in systolic BP (>=30 mmHg) (n=126,124) | 16.7 | 12.9
  Diastolic BP (<50 mmHg) (n=127,127) | 0.8 | 1.6
  Increase in diastolic BP (>=20 mmHg) (n=126,124) | 7.1 | 7.3
  Decrease in diastolic BP (>=20 mmHg) (n=126,124) | 15.9 | 12.9
  Heart rate (>120 bpm) (n=127,127) | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Vital Signs in Cohort 2
Description: Abnormal clinically significant vital signs included absolute systolic BP values: <90 mmHg, maximum increase or decrease of >=30 mmHg from baseline; absolute diastolic BP values: <50 mmHg, maximum increase or decrease of >=20 mmHg from baseline; absolute heart rate values: >120 bpm.
Time Frame: Baseline up to Week 16 (follow-up)
Population: Cohort 2 analysis set included all those participants in the SAS (all participants who receive at least one dose of study medication, including partial doses) who were randomized into cohort 2 of the study. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 2) | Placebo (Cohort 2)
Number analyzed (Participants) | 243 | 244
percentage of participants
  Systolic BP (<90 mmHg) (n=243,244) | 0.8 | 0.0
  Increase in systolic BP (>=30 mmHg) (n=240,240) | 3.8 | 8.3
  Decrease in systolic BP (>=30 mmHg) (n=240,240) | 9.6 | 8.8
  Diastolic BP (<50 mmHg) (n=243,244) | 1.2 | 0.8
  Increase in diastolic BP (>=20 mmHg) (n=240,240) | 6.3 | 5.4
  Decrease in diastolic BP (>=20 mmHg) (n=240,240) | 6.7 | 7.5
  Heart rate (>120 bpm) (n=243,244) | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings in Cohort 1
Description: Abnormal ECG findings included maximum value of >=300 millisecond (msec), maximum increase of >=25% for baseline value of >200 msec and maximum increase of >=50% for baseline value of <=200 msec for PR interval (int); maximum value of >=200 msec, maximum increase of >=25% for baseline value of >100 msec and maximum increase of >=50% for baseline value of <=100 msec for QRS interval; maximum value of >=500 msec for QT interval; maximum value of 450 to <480, 480 to <500 and >=500 msec, increase of >=30 to <60 and >=60 msec for QT interval corrected using Fridericia's formula (QTcF interval).
Time Frame: Baseline up to Week 30 (follow-up)
Population: Cohort 1 analysis set included all those participants in the SAS (all participants who received at least one dose of study medication, including partial doses) who were randomized into cohort 1 of the study. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 1) | Placebo (Cohort 1)
Number analyzed (Participants) | 127 | 127
percentage of participants
  PR int (>=300 msec) (n=123,113) | 0.0 | 0.0
  Increase in PR int (>=25/50%) (n=122,112) | 0.0 | 0.0
  QRS int (>=200 msec) (n=127,127) | 0.0 | 0.0
  Increase in QRS int (>=25/50%) (n=126,126) | 1.6 | 0.0
  QT int (>=500 msec) (n=127,127) | 0.0 | 2.4
  QTcF int (450 to <480 msec) (n=127,127) | 15.7 | 13.4
  QTcF int (480 to <500 msec) (n=127,127) | 1.6 | 4.7
  QTcF int (>=500 msec) (n=127,127) | 0.0 | 0.8
  Increase in QTcF int (>=30 to <60msec )(n=126,126) | 9.5 | 7.1
  Increase in QTcF int (>=60 msec) (n=126,126) | 0.8 | 0.0

4. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings in Cohort 2
Description: Abnormal ECG findings included maximum value of >=300 msec, maximum increase of >=25% for baseline value of >200 msec and maximum increase of >=50% for baseline value of <=200 msec for PR interval; maximum value of >=200 msec, maximum increase of >=25% for baseline value of >100 msec and maximum increase of >=50% for baseline value of <=100 msec for QRS interval; maximum value of >=500 msec for QT interval; maximum value of 450 to <480, 480 to <500 and >=500 msec, increase of >=30 to <60 and >=60 msec for QT interval corrected using Fridericia's formula (QTcF interval).
Time Frame: Baseline up to Week 16 (follow-up)
Population: Cohort 2 analysis set included all those participants in the SAS (all participants who received at least one dose of study medication, including partial doses) who were randomized into cohort 2 of the study. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Groups:
- Dimebon (Cohort 2): Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day up to Week 12.
Arm/Group | Dimebon (Cohort 2) | Placebo (Cohort 2)
Number analyzed (Participants) | 243 | 244
percentage of participants
  PR int (>=300 msec) (n=232,232) | 0.9 | 0.0
  Increase in PR int (>=25/50%) (n=231,229) | 0.0 | 0.0
  QRS int (>=200 msec) (n=243,244) | 0.0 | 0.0
  Increase in QRS int (>=25/50%) (n=242,243) | 0.8 | 0.4
  QT int (>=500 msec) (n=243,244) | 0.8 | 0.8
  QTcF int (450 to <480 msec) (n=243,244) | 15.6 | 19.3
  QTcF int (480 to <500 msec) (n=243,244) | 2.1 | 0.8
  QTcF int (>=500 msec) (n=243,244) | 1.2 | 0.0
  Increase in QTcF int (>=30 to <60 msec)(n=242,243) | 6.6 | 5.8
  Increase in QTcF int (>=60 msec) (n=242,243) | 0.4 | 0.0

5. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Laboratory Values in Cohort 1
Description: For hematology, liver function, renal function, electrolytes, clinical chemistry, abnormality was reported if the observed value was more than or less than X times the upper limit of normal (ULN) or lower limit of normal (LLN) respectively; X=specified in categories of each parameter in the measured values section. For urinalysis of glucose, ketones, protein, blood, abnormality was reported if result was >=1 in qualitative test of respective parameters, indicating levels in urine were abnormal. Urine pH and specific gravity abnormality reported if pH >8 and specific gravity <1.003 or >1.030.
Time Frame: Baseline up to Week 30 (follow-up)
Population: Cohort 1 analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for each group respectively. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 1) | Placebo (Cohort 1)
Number analyzed (Participants) | 126 | 124
percentage of participants
  Hemoglobin (<0.8*LLN) (n=126,123) | 1 | 1
  Red blood cell count (<0.8*LLN) (n=126,123) | 2 | 0
  Mean corpuscular volume (<0.9*LLN) (n=126,123) | 0 | 2
  Mean corpuscular volume (>1.1*ULN) (n=126,123) | 0 | 0
  White blood cell count (<0.6*LLN) (n=126,123) | 0 | 1
  White blood cell count (>1.5*ULN) (n=126,123) | 1 | 0
  Lymphocytes (<0.8*LLN) (n=126,123) | 2 | 1
  Lymphocytes (>1.2*ULN) (n=126,123) | 1 | 2
  Total Neutrophils (<0.8*LLN) (n=126,123) | 0 | 1
  Total Neutrophils (>1.2*ULN) (n=126,123) | 4 | 3
  Monocytes (>1.2*ULN) (n=126,123) | 0 | 1
  Total bilirubin (>1.5*ULN) (n=125,123) | 1 | 2
  Aspartate aminotransferase (>3.0*ULN) (n=125,123) | 1 | 0
  Alanine aminotransferase (>3.0*ULN) (n=125,123) | 1 | 1
  Blood urea nitrogen (>1.3*ULN) (n=125,123) | 1 | 2
  Creatinine (>1.3*ULN) (n=125,123) | 2 | 0
  Sodium (<0.95*LLN) (n=125,123) | 0 | 1
  Sodium (>1.05*ULN) (n=125,123) | 0 | 1
  Potassium (<0.9*LLN) (n=125,123) | 0 | 2
  Potassium (>1.1*ULN) (n=125,123) | 2 | 1
  Calcium (>1.1*ULN) (n=125,123) | 1 | 0
  Magnesium (<0.9*LLN) (n=125,123) | 0 | 0
  Magnesium (>1.1*ULN) (n=125,123) | 20 | 24
  Phosphate (<0.8*LLN) (n=125,123) | 0 | 0
  Phosphate (>1.2*ULN) (n=125,123) | 0 | 0
  Bicarbonate (<0.9*LLN) (n=125,123) | 2 | 0
  Bicarbonate (>1.1*ULN) (n=125,123) | 0 | 1
  Glucose (>1.5*ULN) (n=125,123) | 9 | 10
  Creatine kinase (>2.0*ULN) (n=125,123) | 3 | 2
  Urine specific gravity (<1.003) (n=125,123) | 0 | 0
  Urine specific gravity (>1.030) (n=125,123) | 2 | 2
  Urine pH (>8) (n=125,123) | 0 | 1
  Urine glucose (>=1) (n=125,123) | 4 | 3
  Urine ketones (>=1) (n=125,123) | 1 | 2
  Urine blood (>=1) (n=125,123) | 32 | 7
  Urine protein (>=1) (n=125,123) | 4 | 2

6. Primary Outcome: Percentage of Participants With Abnormal Clinically Significant Laboratory Values in Cohort 2
Description: For hematology, liver function, renal function, electrolytes, clinical chemistry, abnormality was reported if the observed value was more than or less than X times the ULN or LLN respectively; X=specified in categories of each parameter in the measured values section. For urinalysis of glucose, ketones, protein, blood, abnormality was reported if result was >=1 in qualitative test of respective parameters, indicating levels in urine were abnormal. Urine pH and specific gravity abnormality reported if pH >8 and specific gravity <1.003 or >1.030.
Time Frame: Baseline up to Week 16 (follow-up)
Population: Cohort 2 analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure for each group respectively. Here, 'n' signifies those participants who were evaluable for particular category for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 2) | Placebo (Cohort 2)
Number analyzed (Participants) | 239 | 241
percentage of participants
  Hemoglobin (<0.8*LLN) (n=239,241) | 0 | 0
  Red blood cell count (<0.8*LLN) (n=239,241) | 0 | 0
  Mean corpuscular volume (<0.9*LLN) (n=239,241) | 0 | 0
  Mean corpuscular volume (>1.1*ULN) (n=239,241) | 0 | 0
  White blood cell count (<0.6*LLN) (n=239,241) | 0 | 0
  White blood cell count (>1.5*ULN) (n=239,241) | 0 | 0
  Lymphocytes (<0.8*LLN) (n=239,241) | 1 | 0
  Lymphocytes (>1.2*ULN) (n=239,241) | 3 | 0
  Total Neutrophils (<0.8*LLN) (n=239,241) | 0 | 1
  Total Neutrophils (>1.2*ULN) (n=239,241) | 2 | 1
  Monocytes (>1.2*ULN) (n=239,241) | 0 | 0
  Total bilirubin (>1.5*ULN) (n=239,241) | 0 | 0
  Aspartate aminotransferase (>3.0*ULN) (n=239,241) | 0 | 0
  Alanine aminotransferase (>3.0*ULN) (n=239,241) | 0 | 0
  Blood urea nitrogen (>1.3*ULN) ((n=239,241) | 0 | 0
  Creatinine (>1.3*ULN) (n=239,241) | 0 | 1
  Sodium (<0.95*LLN) (n=239,241) | 0 | 0
  Sodium (>1.05*ULN) (n=239,241) | 0 | 0
  Potassium (<0.9*LLN) (n=239,241) | 0 | 0
  Potassium (>1.1*ULN) (n=239,241) | 0 | 0
  Calcium (>1.1*ULN) (n=239,241) | 0 | 0
  Magnesium (<0.9*LLN) (n=239,241) | 0 | 0
  Magnesium (>1.1*ULN) (n=239,241) | 18 | 17
  Phosphate (<0.8*LLN) (n=239,241) | 0 | 0
  Phosphate (>1.2*ULN) (n=239,241) | 0 | 0
  Bicarbonate (<0.9*LLN) (n=239,241) | 0 | 0
  Bicarbonate (>1.1*ULN) (n=239,241) | 0 | 0
  Glucose (>1.5*ULN) (n=239,241) | 6 | 4
  Creatine kinase (>2.0*ULN) (n=239,241) | 3 | 1
  Urine specific gravity (<1.003) (n=237,240) | 0 | 0
  Urine specific gravity (>1.030) (n=237,240) | 2 | 1
  Urine pH (>8) (n=237,240) | 0 | 0
  Urine glucose (>=1) (n=237,240) | 3 | 3
  Urine ketones (>=1) (n=237,240) | 0 | 0
  Urine blood (>=1) (n=237,240) | 26 | 5
  Urine protein (>=1) (n=237,240) | 1 | 3

7. Primary Outcome: Percentage of Participants With Adverse Events (AEs) in Cohort 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 30 (follow-up)
Population: Cohort 1 analysis set included all those participants in the SAS (all participants who received at least one dose of study medication, including partial doses) who were randomized into cohort 1 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 1) | Placebo (Cohort 1)
Number analyzed (Participants) | 127 | 127
percentage of participants | 64.6 | 64.6

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs) in Cohort 2
Description: as for outcome 7
Time Frame: Baseline up to Week 16 (follow-up)
Population: Cohort 2 analysis set included all those participants in the SAS (all participants who received at least one dose of study medication, including partial doses) who were randomized into cohort 2 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Dimebon (Cohort 2) | Placebo (Cohort 2)
Number analyzed (Participants) | 243 | 244
percentage of participants | 55.1 | 53.3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dimebon | Placebo
Serious Adverse Events (participants affected / at risk) | 26/370 | 28/371
Other Adverse Events (participants affected / at risk) | 107/370 | 110/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=370) | Placebo (N=371)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Uterine rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Grand mal convulsion (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Belligerence (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Bladder irritation (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=370) | Placebo (N=371)
Constipation (Gastrointestinal disorders) | 2 | 9
Diarrhoea (Gastrointestinal disorders) | 13 | 9
Nausea (Gastrointestinal disorders) | 8 | 9
Fatigue (General disorders) | 19 | 9
Oedema peripheral (General disorders) | 11 | 9
Urinary tract infection (Infections and infestations) | 26 | 27
Fall (Injury, poisoning and procedural complications) | 15 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Dizziness (Nervous system disorders) | 9 | 9
Headache (Nervous system disorders) | 14 | 10
Somnolence (Nervous system disorders) | 19 | 7
Agitation (Psychiatric disorders) | 8 | 5
Anxiety (Psychiatric disorders) | 3 | 9
Confusional state (Psychiatric disorders) | 4 | 9
Insomnia (Psychiatric disorders) | 5 | 9

LIMITATIONS AND CAVEATS:
This safety study did not specify primary or secondary outcome measures. Relevant summaries of all safety assessments are thus provided. Urine blood abnormalities seen are deemed due to interference with dipstick test by a metabolite of dimebon.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.